CLINICAL TRIAL: NCT06510023
Title: Preserved Reward Sensitivity During Acute Rehabilitation Following Acquired Brain Injury
Brief Title: Rewards Sensitivity After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Shira Cohen-Zimerman, Research Scientist, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: STU00213877
Record Dates: First submitted 2024-07-11; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Acquired Brain Injury
Keywords: Rewards Sensitivity; Motivation; Acquired Brain Injury; Electrodermal Activity
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: 2X3 non-randomized, within-participant design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Acquired Brain Injury (Experimental): Measuring the effect of three different types of rewards (one dollar, one penny, and no reward) on performance in a cognitive test.
  Interventions: Behavioral: Type of reward presented
- Non-impaired controls (Other): Measuring the effect of three different types of rewards (one dollar, one penny, and no reward) on performance in a cognitive test.
  Interventions: Behavioral: Type of reward presented

INTERVENTIONS:
Behavioral: Type of reward presented — Three different types of rewards were presented to both groups during the computerized task: one dollar, one penny, and no reward.

SUMMARY:
A study measuring rewards sensitivity in individuals with acquired brain injury at an acute rehabilitation level.

DETAILED DESCRIPTION:
Individuals in acute rehabilitation following acquired brain injury journal (ABI) and aged-matched, non-injured controls will be recruited for this study.

Testing sessions will take place in a private treatment room at the Shirley Ryan AbilityLab and required 45 minutes to complete. Upon entering the room, participants will be greeted, electrodes placed on the participant's fingers to record their electrodermal activity, and participants will provide demographic information. Participants will then be instructed about how to respond on the Cued Reinforcement Response Time task (CRRT, see description below), and complete the task on a laptop computer while their electrodermal activity is being recorded. In this task, they are instructed to respond as quickly and accurately as possible, and will be informed that they will receive a monetary reward based on their accuracy at the completion of the task. Finally, participants will complete 3 self-report measures: (1) explicit level of motivation was measured in a post-study survey which included two items from the Sensitivity to Punishment and Sensitivity to Reward Questionnaire, (SPSRQ); (2) Reward sensitivity was evaluated using the Reward Responsiveness Scale , and (3) depression was evaluated using the Patient Health Questionnaire (PHQ-8) survey. At the end of the session, the electrodes will be removed, and participants will be debriefed and provided their monetary reward

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ABI

  * Diagnosis of Traumatic Brain Injury or Stroke, based on their medical records
  * Age between 18-100
  * Able to follow directions in English (measured informally during screening)
  * Able to use at least one upper extremity (demonstrated by holding a pen)
  * Mild-moderate or lesser diagnosis in cognitive-communication area
  * Score of 25 or higher on the Orientation Log assessment
  * Able to consent for participation in study (identifies through chart review)
  * Capable of understanding and cooperating with the experimental procedures.

Healthy participants

* Age of 18 to 100 years old
* Ability to follow directions in English
* Ability to use at least one upper extremity.

Exclusion Criteria:

* Individuals with ABI

  * Additional diagnosis of a neurological disorder other than ABI
  * Additional diagnosis of aphasia.
  * Having cognitive or behavioral impairments that preclude participation in the experimental procedures

Healthy Participants

• history of significant cerebrovascular or neurological disease including (but not limited to) meningitis, epilepsy and/or seizures, stroke, tumor, multiple sclerosis, meningitis, mental retardation, dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Performance on a Cued Response Reaction Time Task, in each of the three rewards conditions (Dollar, Penny, No reward) | 15 minutes
  Accuracy (percentage of correct responses) in a Cued Response Reaction task
Performance on a Cued Response Reaction Time Task, in each of the three rewards conditions (Dollar, Penny, No reward) | 15 minutes
  Response time (time in milliseconds) in a Cued Response Reaction task
Electrodermal activity (EDA) before, during and after the Cued Response Reaction task | 30 minutes
  Number of skin conductance responses (SCRs) before, during and after the task

CONTACTS AND LOCATIONS:
Overall Officials: Shira Cohen-Zimerman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No